CLINICAL TRIAL: NCT01425710
Title: Non-invasive Evaluation of Fluid Status and Cardiac Output During Operative Treatment of Pheochromcytoma
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martin Niederle, MD, DMedSc, Medical University of Vienna
Other Study IDs: pheo
Record Dates: First submitted 2011-08-24; First posted 2011-08-30 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pheochromocytoma
Keywords: Pheochromocytoma; Adrenalectomy; Cardiac output; Fluid managment; Esopagheal doppler sonography
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pheochromocytoma Group: Intraoperative esophageal doppler sonography during laparoscopic adrenalectomy performed for pheochromocytoma
- Control group: Intraoperative esophageal doppler sonography during laparoscopic adrenalectomy for non-pheochromocytoma adrenal tumor

SUMMARY:
Non-invasive measurements of cardiac output (CO), systemic vascular resistance (SVR), corrected aortic flow time (FTc) and stroke volume (SV) are useful parameters during laparoscopic resection of pheochromocytoma (adrenalectomy) to document the intraoperative changes in volume status and to estimate the volume depletion.

DETAILED DESCRIPTION:
Pheochromocytomas and extraadrenal paragangliomas are catecholamin-producing tumours deriving from the adrenal medulla and sympathetic ganglia. The only causal therapy is surgical resection. Nowadays, laparoscopic adrenalectomy is thought to be the optimal approach. Chronic volume depletion due to chronic hypertension and preoperative α-adrenoreceptor-blockade (to avoid the effects of intraoperative catecholamine-excess) often lead to hypotension after resection of the tumour. Volume reload with high amounts of fluid is often needed. Therefor some authors recommended invasive measurement (pulmonary artery catheter) to control cardiac output parameters and fluid balance. However, there are non-invasive methods to measure cardiac output(CO), systemic vascular resistance(SVR), stroke volume(SV) and corrected aortic flow time(FTc) to estimate volume status. Except transesophageal echocardiography, other techniques such as transoesophageal doppler and pulse pressure methods exist but have not been investigated during surgical therapy for pheochromocytoma so far. The esophageal Doppler currently represents the "gold standard" for perioperative fluid replacement therapy.

The study's hypothesis is that non-invasive measurements of cardiac output (CO), systemic vascular resistance (SVR), corrected aortic flow time (FTc) and stroke volume (SV) are useful parameters during laparoscopic resection of pheochromocytoma (adrenalectomy) to document the intraoperative changes in volume status and to estimate the volume depletion.

ELIGIBILITY:
Inclusion Criteria:

* Planned laparoscopic adrenalectomy for pheochromocytoma (Biochemical confirmed adrenal and extraadrenal pheochromocytoma)
* Planned laparoscopic adrenalectomy for hormonally inactive adrenal tumor

Exclusion Criteria:

* Risk of esophageal bleeding or perforation exists (i.e., liver disease with portal hypertension and/or esophageal varicoses, other esophageal anomalies).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from pheochromocytoma will be recruited by the Department of Surgery, Medical University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output (CO) | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  measured using esophageal doppler
Systemic vascular resistance (SVR) | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  measured using esophageal doppler
Stroke volume (SV) | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  measured using esophageal doppler
Corrected aortic flow time(FTc) | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  measured using esophageal doppler
Central venous pressure | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  Measured using esophageal doppler
Heart rate | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
Arterial blood pressure | parameter will be measured continously for the duration of adrenalectomy, an expected average of 3 hours
  systolic, diastolic, mean; continuous invasive measurement

SECONDARY OUTCOMES:
Changes in serum Concentration: Epinephrine | 7 timepoints during anesthesia (Administration of rocuronium, intubation, cut, intraabdominal air insufflation, ligature of v. suprarenalis, tumor exstirpation, end of operation)
Changes in serum concentration: Norepinephrine | 7 timepoints during anesthesia (Administration of rocuronium, intubation, cut, intraabdominal air insufflation, ligature of v. suprarenalis, tumor exstirpation, end of operation)
Changes in serum concentration: Dopamin | 7 timepoints during anesthesia (Administration of rocuronium, intubation, cut, intraabdominal air insufflation, ligature of v. suprarenalis, tumor exstirpation, end of operation)
Changes in plasma concentration: Metanephrines | 7 timepoints during anesthesia (Administration of rocuronium, intubation, cut, intraabdominal air insufflation, ligature of v. suprarenalis, tumor exstirpation, end of operation)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Niederle, MD, DMedSc, Principal Investigator — Medical University of Vienna; Edith Fleischmann, Prof, MD, Study Chair — Medical University of Vienna; Bruno Niederle, Prof, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Niederle MB, Fleischmann E, Kabon B, Niederle B. The determination of real fluid requirements in laparoscopic resection of pheochromocytoma using minimally invasive hemodynamic monitoring: a prospectively designed trial. Surg Endosc. 2020 Jan;34(1):368-376. doi: 10.1007/s00464-019-06777-z. Epub 2019 Apr 11. PMID 30976898